CLINICAL TRIAL: NCT02839525
Title: The Effect of Nutritional Interventions on Exercise-induced Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Letícia Chisini Loss, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 51384015.5.0000.5345
Record Dates: First submitted 2016-07-13; First posted 2016-07-21 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Muscle Damage
Keywords: Eccentric exercise; Dietary supplement; Muscle damage
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Omega 3 (Placebo Comparator): * 3000mg of olive oil
  * Eccentric exercise: 100 maximal eccentric contractions of knee extensors, divided into 10 sets of 10 repetitions at intervals of 60 seconds between the series
  Interventions: Dietary Supplement: Omega 3; Other: Eccentric exercise
- Isolate whey protein (Placebo Comparator): * 23g of maltodextrin
  * Eccentric exercise: 100 maximal eccentric contractions of knee extensors, divided into 10 sets of 10 repetitions at intervals of 60 seconds between the series
  Interventions: Dietary Supplement: Isolate whey protein; Other: Eccentric exercise
- Omega 3 and Isolate whey protein (Placebo Comparator): * 3000mg of olive oil and 23g of maltodextrin
  * Eccentric exercise: 100 maximal eccentric contractions of knee extensors, divided into 10 sets of 10 repetitions at intervals of 60 seconds between the series
  Interventions: Dietary Supplement: Omega 3 and Isolate whey protein; Other: Eccentric exercise

INTERVENTIONS:
Dietary Supplement: Omega 3 — 3000mg of n-3 oil (2000mg EPA e 1000mg DHA)
  Arms: Omega 3
Dietary Supplement: Isolate whey protein — 23g of protein of whey protein
  Arms: Isolate whey protein
Dietary Supplement: Omega 3 and Isolate whey protein — 3000mg of n-3 oil (2000mg EPA e 1000mg DHA) and 23g of protein of whey protein
  Arms: Omega 3 and Isolate whey protein
Other: Eccentric exercise — 100 maximal eccentric contractions of knee extensors, divided into 10 sets of 10 repetitions at intervals of 60 seconds between the series

SUMMARY:
The study is a randomized, double-blinded, placebo-controlled trial that will include the participation of 69 women, aged 18-40 years. The aim of the study is to test nutritional strategies that help to minimize the effects of muscle damage induced by exercise.

The procedures will be performed at the Federal University of Health of Porto Alegre (UFCSPA).

DETAILED DESCRIPTION:
The exercise-induced muscle damage is associated with eccentric activities affecting muscle structural unit through micro-injury that can promote a local inflammatory response, muscle damage and delayed onset muscle soreness. These events can cause an impact on athletic performance and lower adherence to the training programs. To optimize muscle recovery after the damage caused by exercise is essential to ensure adequate caloric intake , with required amounts of macronutrients and micronutrients. Recent studies have been showed that the protein intake before sleeping is a effective strategy to inhibit muscle protein degradation, stimulate muscle protein synthesis and facilitate adaptive response of skeletal muscle to physical exercise. Furthermore, evidences on the use of anti-inflammatory nutrients have suggested that diets rich in omega 3 can reduce inflammation through inhibition of pro-inflammatory mediators. Therefore, the intake of this nutrient combined with a protein meal before sleeps and the control of food intake can improve adherence to sports training. The study will consist of three groups where everyone will receive an individualized diet. A randomization procedure will determine the type of intervention. The distribution of the groups will be as follows: group 1 (control) - volunteers follow individualized diet and olive oil capsules and maltodextrin; group 2 - intervention with omega 3 more individualized diet ; group 3 - omega 3 and whey protein isolate intervention more individualized diet.

The order of procedures to be performed will be: (1) Nutritional and Anthropometric assessment; (2) Individual orientation of diet and distribution of supplements; (3) Baseline assessment (peak torque, muscle pain levels and vastus lateralis and rectus femoris echo intensity; (4) Muscle damage induction by eccentric exercise protocol; (5) Reviews after 24h, 48h, 72h, which will follow the routine and the methods applied at baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 years aged
* BMI 18,5-25kg/m2
* physical exercise: < 150 minutes per week

Exclusion Criteria:

* pregnancy/ lactation
* vegetarian/vegan
* chronic disease
* pulmonary and neurologic disease
* muscle injury/knee muscle injury
* medication use: anti-inflammatory and anticoagulant
* fish oil and derivate allergy
* dietary supplements use in the last month: whey protein, casein, albumin, glutamin, meat and soy protein, creatine, branched chain amino acid, high calorie supplement, n-3 supplement and antioxidants

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle strength evaluation (Peak Torque) | One Year
  Three maximal isometric contractions of knee extensors will be performed by the isokinetic dynamometer equipment Biodex System 4 Pro (Biodex Medical Systems, USA).

SECONDARY OUTCOMES:
Evaluation of quadriceps muscle pain (Muscle pain levels) | One year
  The assessment of pain as muscle damage marker is expressed by a visual analog scale.
Vastus lateralis and rectus femoris echo intensity | One year
  Ultrasound images

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Dornelles Schneider, Doctor, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- UFCSPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes